CLINICAL TRIAL: NCT03101852
Title: Effectiveness and Acceptability of Nutritional Rehabilitation Based on Ready-to-use Food in HIV-infected Children and Adolescents in Senegal: The Multicentre SNAC'S Study
Brief Title: Nutritional Rehabilitation in Senegalese HIV-infected Children and Adolescents
Acronym: SNAC'S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Global Fund (Other); Sidaction (Other); UNICEF (Other); United Nations World Food Programme (WFP) (Other)
Responsible Party: Principal Investigator, Cecile Cames, Principal investigator, Researcher, Institut de Recherche pour le Developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14SANIN203
Record Dates: First submitted 2017-03-22; First posted 2017-04-05 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Malnutrition; HIV/AIDS
Keywords: severe acute malnutrition; moderate acute malnutrition; HIV-infection; adolescents; antiretroviral; Africa; ready-to-use food; outpatient care
MeSH Terms: conditions — Malnutrition; Acquired Immunodeficiency Syndrome; Severe Acute Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional therapy (Experimental): Children included in the study with severe acute malnutrition receive Plumpy Nut: WHO recommends a Plumpy Nut® prescription of 75 to 100 kcal/kg/d in children aged 5 to 10 years and 60 to 90 kcal/kg/d above that age. The lowest value was used and maximum energy intake provided by RUF was limited to 2,000 kcal/d i.e. 4 sachets in order to preserve habitual diet and prevent appetite saturation
  Interventions: Dietary Supplement: Plumpy Nut
- Nutritional supplementation (Experimental): Children included in the study with moderate acute malnutrition receive Plumpy Sup: 60kcal/kg/day, limited to 4 doses/day.
  Interventions: Dietary Supplement: Plumpy Sup

INTERVENTIONS:
Dietary Supplement: Plumpy Nut
  Other Names: ready-to-use therapeutic food
  Arms: Nutritional therapy
Dietary Supplement: Plumpy Sup
  Other Names: ready-to-use supplementary food
  Arms: Nutritional supplementation

SUMMARY:
Severe (SAM, Body Mass Index-z < -3) and moderate (MAM, -3 ≤ BMI-z < -2) acute malnutrition, highly prevalent in HIV-infected children and adolescents, is an independent risk factor of death, even when antiretroviral treatment (ART) is initiated. The objectives of the SNAC'S study are to assess acceptability and effectiveness of outpatient nutritional rehabilitation, using ready-to-use food (RUF), elaborated in compliance with national and international recommendations and implemented in HIV-infected children and adolescents, under active follow-up in the 12 main pediatric HIV care sites in Senegal and presenting with SAM or MAM.

DETAILED DESCRIPTION:
Background:

Severe (SAM, BMI-z < -3) and moderate (MAM, -3 ≤ BMI-z < -2) acute malnutrition, highly prevalent in HIV-infected children and adolescents, is an independent risk factor of death, even when antiretroviral treatment (ART) is initiated. Scaling-up of ART decreased morbimortality in children in low-income settings and thus allowed HIV-infection to become, to some extent, a chronic disease. However, appropriate and targeted nutritional interventions take a long time to be assessed with the aim of their integration in the "global care" of HIV infection, thus jeopardizing in these patients who go through adolescence the successes achieved so far. Many clinical trials reported a greater efficacy of the ready-to-use therapeutic foods (RUTF) in the nutritional rehabilitation compared with standard interventions, among up to five children, with or without HIV-infection. Since 2007, the United Nations recommend their use for the outpatient nutritional rehabilitation of severely malnourished children and since 2009, also in HIV-infected adolescents.

Objectives :

The objectives of the SNAC'S study are to assess acceptability and effectiveness of outpatient nutritional rehabilitation, using ready-to-use food (RUF), elaborated in compliance with national and international recommendations and implemented in HIV-infected children and adolescents, under active follow-up in the 12 main pediatric HIV care sites in Senegal.

Will be specifically assessed:

Effectiveness of nutritional rehabilitation in terms of catch-up weight growth, of immunologic status improvements, of muscular mass gain and of micronutrients status (including the correlation within these outcomes). Long-term (3 months and 6 months after discharge) weight growth and relapse will be assessed Acceptability of the intervention will be assessed using quantitative methods (observance to RUF prescription, feeding modalities, organoleptic appreciation, etc.) and qualitative methods (focus group and interviews about perceptions among children > 7 years and health workers).

The SNACS study was carried out in Senegal from April 2015 to January 2017 in 12 public paediatric clinics: two in the Dakar district, the capital city, (Albert Royer National Paediatric Hospital and Roi Baudouin Hospital) and 10 in decentralized settings (Regional Hospitals of Saint Louis, Louga, Mbour, Kaoloack, Ziguinchor and Kolda; Health centres of Thiès, Nioro du Rip, Bignona and Kolda). Study implementation was gradual, starting with the central sites in April 2015 and ending with the Kolda sites in March 2016.

Methods:

This is an open cohort study (intervention/evaluation) conducted over 2 years. Children with SAM will be enrolled in a rehabilitation protocol, using Plumpy Nut until the target weight is reached, BMI-z > -2. Children with MAM will be enrolled in a rehabilitation protocol, using Plumpy Sup. At enrollment and at discharge from the rehabilitation protocols, a blood sample will be collected for an immunovirological, biological and selected proteins and micronutrients assessment. At each visit, a clinical examination and anthropometric measurements will be performed.

At enrollment and after discharge, focus groups will be conducted with children > 7 years about their understanding and perception of the study protocol and of the nutritional care. Before enrollments start and at the end of the study, interviews will be conducted with the health workers involved in the study to explore their understanding of the study and their perceptions about the acceptability, effectiveness and feasibility of the nutritional rehabilitation of HIV children. Overall acceptability of RUF will be assessed in children by questionnaires at 3 time points during the study follow-up.

Expected outcomes:

Implementation of the recent recommendations on early ART initiation in children should allow the integration of targeted and appropriate nutritional interventions. The SNAC's Study will disseminate the first scientific data on modalities, acceptability and efficacy of nutritional rehabilitation in HIV-infected older children and adolescents in Africa. As it complies with international and national recommendations, it will also provide programmatic data, with regards to feasibility of outpatient nutritional rehabilitation using RUTF in HIV-infected adolescents, to national stakeholders and decision makers. It is ultimately expected to facilitate effective integration of these vulnerable patients both in nutritional care guidelines and follow-up health structures.

ELIGIBILITY:
Inclusion Criteria:

* infected with HIV
* presenting with severe or moderate acute malnutrition
* followed-up in one of the 12 study sites
* written consent of the parent/legal guardian
* verbal assent of the child

Exclusion Criteria:

* pregnancy
* physical and/or mental disability incompatible with the study follow-up
* living far from the study site (about more than 50km)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 185 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Successful nutritional rehabilitation | up to 12 months
  the child reach his/her target weight defined as weight-for-height >= - 2 z-scores in children < 5years; body mass index for age >= -2 z-score in children >= 5 years

SECONDARY OUTCOMES:
long-term effectiveness | 3 months
  the child maintains stable weight (or gains weight) 3 months after reaching target weight.
long-term effectiveness | 6 months
  the child maintains stable weight (or gains weight) 6 months after reaching target weight.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Diop, MD, Principal Investigator — Division de Lutte contre le Sida et les IST, Dakar, Senegal; Fatou Niasse-Traore, MD, Principal Investigator — Comité National de Lutte contre le Sida, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Niasse F, Varloteaux M, Diop K, Ndiaye SM, Diouf FN, Mbodj PB, Niang B, Diack A, Cames C. Adherence to ready-to-use food and acceptability of outpatient nutritional therapy in HIV-infected undernourished Senegalese adolescents: research-based recommendations for routine care. BMC Public Health. 2020 May 15;20(1):695. doi: 10.1186/s12889-020-08798-z. PMID 32414346
- [Derived] Hejoaka F, Varloteaux M, Desclaux-Sall C, Ndiaye SM, Diop K, Diack A, Niasse F, Cames C. Improving the informed consent process among HIV-infected undisclosed minors participating in a biomedical research: insights from the multicentre nutritional SNACS study in Senegal. Trop Med Int Health. 2019 Mar;24(3):294-303. doi: 10.1111/tmi.13202. Epub 2019 Jan 24. PMID 30624827